CLINICAL TRIAL: NCT04436380
Title: Retrospective Study of Patients With Severe Aplastic Anemia Who Relapsed After Immunosuppressive Therapy
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999920119; 20-H-N119
Record Dates: First submitted 2020-06-17; First posted 2020-06-18 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Severe Aplastic Anemia
Keywords: Alemtuzumab; rATG; Natural History
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Relapsed SAA Patients: Patients with Severe Aplastic Anemia who Relapsed after Immunosuppressive Therapy

SUMMARY:
Background:

Severe aplastic anemia (SAA) is a form of bone marrow failure. It usually results from a

cytotoxic T cell attack on the marrow stem cell. Two treatments can be used for most people with SAA. One is allogeneic hematopoietic stem cell transplant (HSCT). The other is immunosuppressive treatment (IST). For people who are treated with IST, relapse can occur. If this happens, they can have HSCT or be re-treated with IST. The two most common IST regimes used for relapsed SAA are rabbit ATG (rATG) and alemtuzumab. Both rATG and alemtuzumab have similar response rates and survival rates. There is not much long-term data on people who need repeat IST treatment due to relapse. Researchers want to look at data from past studies to learn more.

Objective:

To compare the data of relapsed SAA patients between those who received alemtuzumab versus rATG for repeat IST treatment.

Eligibility:

Adults and children with SAA who were enrolled on NHLBI protocol 12-H-0150, 06-H-0034, 05-H-0242, 03-H-0249, 03-H-0193, 00-H-0032, or 90-H-0146

Design:

This study uses data from past studies. The participants in those studies have allowed their data to be used in future research.

Researchers will review participants medical records. They will collect clinical data, such as notes, test results, and imaging scans. They will also collect the research data gathered as part of the original study.

Researchers will enter the data into an in-house database. It is password protected. All data will be kept in secure network drives or in secure sites.

Other studies may be added in the future....

DETAILED DESCRIPTION:
Severe aplastic anemia (SAA) is a form of bone marrow failure and in most cases is the result of a cytotoxic T cell attack on the marrow stem cell. It is effectively treated in most patients with either immunosuppressive treatment (IST) or upfront allogeneic hematopoietic stem cell transplant (HSCT). However, in patients who are treated with IST, relapse remains an issue with a rate of 30-40%. Once relapsed, patients can be either re-treated with IST or undergo HSCT. The two most common IST regimes used for relapsed SAA are rabbit ATG (rATG) and alemtuzumab. Both rATG and alemtuzumab have been shown to have a response rate of approximately 60% in relapsed patients with similar overall survival rates of 83-85%. Previous predictors of relapse include time from diagnosis to IST, and early response to IST. Few long-term data exist on patients requiring repeat IST treatment due to relapse.

ELIGIBILITY:
* This is a retrospective chart review. The investigators will review the medical records of adults and children with severe aplastic anemia (SAA) enrolled on immunosuppressive therapy (IST) treatment protocols in the NHLBI.

Patients who opted out of future use of data on their prior studies will be excluded from this study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Relapsed SAA Subjects who had a repeat IST
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Assessment of long-term outcomes of relapsed patients who received repeat IST | Between the Period of 1990 to 2020
  Characteristics and outcomes of relapsed SAA patients between those who received alemtuzumab versus rATG for repeat IST

SECONDARY OUTCOMES:
Clinical predictors for the development of relapse | Between the Period of 1990 to 2020
  Clinical predictors for the development of relapse such as age, gender, baseline laboratory values, time from diagnosis to initial treatment, and initial treatment received.
Rates of clonal evolution between relapsed patients depending on type of IST received and number of IST rounds required | Between the Period of 1990 to 2020
  Compare rates of clonal evolution between relapsed patients depending on type of IST received and number of IST rounds required.

CONTACTS AND LOCATIONS:
Overall Officials: Emma M Groarke, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States